CLINICAL TRIAL: NCT04503135
Title: Prospective Cohort Study on Catheter Associated Asymptomatic Thrombosis in Intensive Care Unit
Brief Title: Catheter Associated Asymptomatic Thrombosis in Intensive Care Unit
Acronym: CAAT
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Mauro Panigada, Principal Investigator, Policlinico Hospital
Other Study IDs: 172_2020
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Central Venous Catheters; Central Venous Catheter Thrombosis; Thrombosis, Venous; Intensive Care Unit
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis; Venous Thrombosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — ultrasound of the central veins of the neck and chest and a (compression ultra-sound) CUS of the femoral veins will be performed bilaterally

SUMMARY:
This study aims to describe the incidence of catheter-related and non-catheter-related thrombosis in a population of adults in ICU and to assess its correlation with alteration of coagulation parameters.

DETAILED DESCRIPTION:
Central venous catheter (CVC) is now indispensable in the monitoring and care of patients in intensive care (ICU). Unfortunately, one of the complications of its positioning is catheter-related thrombosis (CRT) and its consequences. Despite the widespread use of CVC and the extensive literature describing its complications, areas of uncertainty regarding the onset, treatment and prevention of CRT persist, especially with regard to asymptomatic thrombosis.

This study aims to describe the incidence of catheter-related and non-catheter-related thrombosis in a population of adults in ICU and to assess its correlation with alteration of coagulation parameters.

The main objective of this study is to assess the proportion of patients developing CRT (proportion) and the incidence of CRT (rate expressed in catheter events/days) in patients in ICU.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18
* admitted to intensive care who have for clinical reasons need to place a central venous catheter
* signing of informed consent

Exclusion Criteria:

* patients under 18 years of age
* Known cancer status
* Congenital thrombophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Unit (ICU) adult patients requiring Central venous catheter for clinical reasons
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Proportion of patients developing Catheter related thrombosis and Incidence of CRT in patients in ICU | Until CVC removal
  The main objective of this study is to assess the proportion of patients developing CRT (proportion) and the incidence of CRT (rate expressed in catheter events/days) in patients in ICU.

SECONDARY OUTCOMES:
Proportion of various types of thrombotic apposition | Until CVC removal
  The proportion of various types of thrombotic apposition
Deep venous thrombosis (DVT) proportion and Incidence | Until CVC removal
  The proportion of patients developing DVT and the incidence of catheter-related DVT (rate) in patients in ICU carrying CVC.
the association of thrombosis with alterations of hemocoagulative parameters | Until CVC removal
  the association of thrombosis with alterations of hemocoagulative parameters
describe the clinical measures that have been taken following the diagnosis of CRT.describe the clinical measures that have been taken following the diagnosis of CRT. | Until CVC removal
  describe the clinical measures that have been taken following the diagnosis of CRT.

CONTACTS AND LOCATIONS:
Overall Officials: chiara Abbruzzese, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Forauer AR, Theoharis CG, Dasika NL. Jugular vein catheter placement: histologic features and development of catheter-related (fibrin) sheaths in a swine model. Radiology. 2006 Aug;240(2):427-34. doi: 10.1148/radiol.2402031129. PMID 16864670
- [Background] Rooden CJ, Tesselaar ME, Osanto S, Rosendaal FR, Huisman MV. Deep vein thrombosis associated with central venous catheters - a review. J Thromb Haemost. 2005 Nov;3(11):2409-19. doi: 10.1111/j.1538-7836.2005.01398.x. Epub 2005 Jun 24. No abstract available. PMID 15975139
- [Background] Bates SM, Jaeschke R, Stevens SM, Goodacre S, Wells PS, Stevenson MD, Kearon C, Schunemann HJ, Crowther M, Pauker SG, Makdissi R, Guyatt GH. Diagnosis of DVT: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e351S-e418S. doi: 10.1378/chest.11-2299. PMID 22315267
- [Background] Hrdy O, Strazevska E, Suk P, Vach R, Karlik R, Jarkovsky J, Sas I, Gal R. Central venous catheter-related thrombosis in intensive care patients - incidence and risk factors: A prospective observational study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2017 Dec;161(4):369-373. doi: 10.5507/bp.2017.034. Epub 2017 Aug 24. PMID 28839334
- [Background] Nm Bhat M, Venkataraman R, Ramakrishnan N, K Abraham B, Rajagopalan S. Value of Routine Sonographic Screening of Internal Jugular Vein to Detect Catheter Related Thrombosis in Intensive Care Unit. Indian J Crit Care Med. 2019 Jul;23(7):326-328. doi: 10.5005/jp-journals-10071-23207. PMID 31406439